CLINICAL TRIAL: NCT01382875
Title: Medico-social Impact of a Comprehensive Multi-disciplinary Program for the Care of Fragility Fracture of the Elderly -Implications for Healthcare Policy in Hong Kong
Brief Title: The Comparison of Comprehensive Multi-disciplinary Program and Conventional Care Program on Fragility Fracture Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok-Sui Leung, Chair Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 4013-PPR-09
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Hip Fracture
Keywords: Multi-disciplinary management program; Conventional care program; Balance Ability; Quality of Life
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional care program (No Intervention)
- Multi-disciplinary management program (Experimental)
  Interventions: Other: Multi-disciplinary management program

INTERVENTIONS:
Other: Multi-disciplinary management program — conventional healthcare program for fragility fracture patients plus vibration treatment, exercise class and educational talk
  Arms: Multi-disciplinary management program

SUMMARY:
Fragility fractures are one of the commonest injuries among elderly people in Hong Kong and account for 12% of the disease burden in elderly aged 65 or above.

A good management healthcare program and training helps elderly to restore full functional level and prevent re-fracture in the following 2 years after primary fracture, but Hong Kong lacks of such program. Some reports from other countries pointed out a well-organized multi-disciplinary management programs are cost-effective to identify and treat osteoporosis, reduce the fracture rate, improve quality of life and raise awareness of fragility fracture.

This study aims to compare the cost-effectiveness of multi-disciplinary management program with conventional care controls. The clinical effectiveness outcomes (re-fracture rate, fall rate, mortality, mobility, quality of life and specialist follow-up time) of the fragility hip fracture patients in New Territories East receiving the proposed management program will be compared with those from Kowloon Central with usual care as controls. The findings will provide useful data for the policy maker to evaluate the current clinical service for fragility fracture patients and consider the implementation of new multi-disciplinary management program into our healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Fragility hip fracture patients within age 65-90

Exclusion Criteria:

* Taking medication affecting bone metabolism or intensive exercise training;
* Those living in old age homes or anyone who is not able to comply with our program

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cost effectiveness of the multi-disciplinary management program and conventional care program | 1 year
  The expected costs of fragility fracture treatment and re-fracture at the hip are calculated from the prospective of hospital and community center cost, with a time frame of one year.

SECONDARY OUTCOMES:
Mobility | 1 year
  The patients will be asked to perform mobility assessments according to our established protocol, including timed-up-to-go, mobility score, Berg balance scale and fall risk screening. The result of the above assessments will be reported as a scoring to show the level of fall risk of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Kwok-Sui Leung, MD, Principal Investigator — Department of Orthopaedics and Traumatology, The Chinese University of Hong Kong
Locations (1):
- Department of Orthopaedics and Traumatology, The Chinese University of Hong Kong, Hong Kong, China